CLINICAL TRIAL: NCT00440804
Title: Randomized, Double-Blind Study of Ibuprofen L-Lysine Intravenous Solution in Premature Infants for the Early Treatment of Patent Ductus Arteriosus
Brief Title: Safety and Efficacy Study of Ibuprofen l-Lysine Solution in Premature Infants for Treatment of PDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Farmacon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FCR-00-01/CB88
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Patent Ductus Arteriosus
Keywords: patent ductus arterious
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ibuprofen l-lysine iv solution (NeoProfen (R) )

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of ibuprofen l-lysine iv in premature infants in the early treatment of Patent Ductus Arteriosus.

DETAILED DESCRIPTION:
The ductus arteriosus remains patent in about 40% to 80% of very low birth weight infants. Early treatment by intravenous ibuprofen L-lysine (IV ibuprofen) has been suggested in preliminary studies to close the ductus and shorten hospital stay. This study aims to determine the effect of early treatment with IV ibuprofen given to the very low birth weight infant with a non-symptomatic patent ductus arteriosus (PDA) at less than 72 hours of life to accelerate and maintain ductal closure, thereby reducing the need for rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn infant of either gender with a birth weight of 500 to 1000 grams, appropriate for gestational age;
* Non-symptomatic PDA with evidence of ductal shunting documented by an echocardiogram (ECHO);
* Less than 72 hours of age at the time of randomization;
* If infant is one of a multiple birth, he/she is one of the two (2) oldest infants who meet the eligibility criteria;
* Consent form signed by parent.

Exclusion Criteria:

* Either major congenital malformations and/or chromosomal anomalies;
* Proven, severe congenital bacterial infection;
* Maternal antenatal nonsteroidal anti-inflammatory drug (NSAID) exposure < 72 hours prior to delivery;
* Treatment with pharmacological replacement steroid therapy at anytime since birth;
* Unremitting shock requiring very high doses of vasopressors (i.e. inability to maintain mean arterial blood pressure appropriate for gestational age ± 2 SD using volume and maximal vasopressor therapy as defined by the individual institution);
* Renal failure or oliguria defined as urine flow rate < 0.5 mL/kg/hr in the 8 hours prior to randomization (Anuria is acceptable if infant is in first 24 hours of life);
* Platelet count < 75,000/mm 3;
* Clinical bleeding tendency (i.e. oozing from puncture sites);
* Expected survival less than 48 hours in the opinion of the attending neonatologist;
* Participation in other clinical intervention trials. Exceptions may be made if approved by Medical Director or designee, RPD Pharmaceutical Department;
* Symptomatic PDA as documented by 3 of the following 5 criteria
* Bounding pulse
* Hyperdynamic precordium
* Pulmonary edema
* Increased cardiac silhouette
* Systolic murmur Or, in view of the neonatologist is deemed to have a hemodynamically significant ductus.
* Exposure to NSAIDs at any time since birth.

Ages: 28 Weeks to 34 Weeks | Sex: All
Age Groups: Child
Dates: Start 2002-12; Study Completion 2005-08

PRIMARY OUTCOMES:
Primary Outcome Measures (Efficacy)

SECONDARY OUTCOMES:
Gastrointestinal function
Renal function
Hematology
Liver enzyme tests
Serum bilirubin
Respiratory function
Intraventricular hemorrhage
Pulmonary hemorrhage
Pulmonary hypertension
Exploratory outcomes:
Ibuprofen concentrations
Prostanoid concentrations
CYP2C9 Genotyping
Follow-up Outcomes
Retinopathy of Prematurity
Bronchopulmonary dysplsia
Periventricular leukomalacia

CONTACTS AND LOCATIONS:
Overall Officials: Jacob V Aranda, MD, PhD, Principal Investigator